CLINICAL TRIAL: NCT02889887
Title: The Investigation of Relationship Between Sensory Processing and Motor Development in Preterm Infants
Brief Title: Relationship Between Sensory Processing and Motor Development
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Celik, research assistant, Gazi University
Other Study IDs: HalilÇ
Record Dates: First submitted 2016-08-22; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Sensation Disorders
Keywords: Preterm; Sensory Processing; Motor Development
MeSH Terms: conditions — Sensation Disorders; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- preterm: infants who born before 37 completed weeks

SUMMARY:
The aim of this study is to analyse correlation between the sensory processing and motor development in preterm infants.

DETAILED DESCRIPTION:
The aim of this study is to analyse correlation between the sensory processing and motor development in preterm infants. A total of 60 infants who were born preterm (n=30) and term (n=30), the corrected and chronological ages between 10-12 months, were included in this study. Test of Sensory Function in Infants was used to evaluate sensory processing, and Alberta Infant Motor Scale was used to evaluate motor development.Spearman correlation test indicated strong positive relation between sensory processing and motor development in preterm infants. Given the relationship between sensory processing and motor development in preterm group, for effective implementation of physiotherapy assessments and interventions, it was thought that it is necessary to evaluate the sensory processing as well as the motor development in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* gestational age lower than 37 month
* corrected age within 10-12 months
* without congenital anomaly or systemic disease
* stay in Neonatal Intensive Care Unit (NICU) at least 2 weeks

Exclusion Criteria:

* taken physiotherapy or sensory integration therapy in any rehabilitation center
* having newborn retinopathy

Ages: 10 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 60 infants who were born preterm (n=30) and term (n=30), the corrected and chronological ages between 10-12 months, were included in this study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The investigation of sensory processing in preterm infants | Day 1
  Test of Sensory Function in Infants' was used to evaluate sensory processing in preterm infants.

SECONDARY OUTCOMES:
The investigation of motor development in preterm infants | Day 1
  Alberta Infant Motor Scale' was used to evaluate motor development in preterm infants.

CONTACTS AND LOCATIONS:
Overall Officials: HALİL İ ÇELİK, Principal Investigator — Gazi University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celik HI, Elbasan B, Gucuyener K, Kayihan H, Huri M. Investigation of the Relationship Between Sensory Processing and Motor Development in Preterm Infants. Am J Occup Ther. 2018 Jan/Feb;72(1):7201195020p1-7201195020p7. doi: 10.5014/ajot.2018.026260. PMID 29280716